CLINICAL TRIAL: NCT02833922
Title: Perfect- and Typical-use Effectiveness of the Dot Fertility App Over 13 Cycles: Results From a Prospective Contraceptive Effectiveness Trial
Brief Title: Effectiveness and Efficacy of Dynamic Optimal Timing, a Smart Phone App for Avoiding Pregnancy: an Observational Study
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: Cycle Technologies (Industry); EastBanc Technologies (Industry)
Responsible Party: Principal Investigator, Victoria Jennings, PhD, Director, Georgetown University
Other Study IDs: GR409775
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Desire to Avoid Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women using Dot to avoid pregnancy: Women living in the United States, ages 18-39 who have not used hormonal birth control or been pregnant in the last three months, who are in a relationship with a male sexual partner, and who wish to use the Dot app to avoid pregnancy for at least one year.
  Interventions: Behavioral: Women using Dot to avoid pregnancy

INTERVENTIONS:
Behavioral: Women using Dot to avoid pregnancy — Women who have chosen to use Dot to prevent pregnancy will be followed for 13 cycles to assess perfect and typical use of the Dynamic Optimal Timing method.

SUMMARY:
The purpose of this study is to assess the effectiveness and efficacy of Dynamic Optimal Timing (DOT), an app-based method of family planning that can be used via Android devices, for women who use the method to avoid pregnancy.

DETAILED DESCRIPTION:
This is a prospective, efficacy study of the Dynamic Optimal Timing (Dot), an app-based method of family planning that provides the user with information about her daily probability of pregnancy based on the length of her menstrual cycles over time. To use the app, women enter the first day of their menstrual period. Women are then provided information about their daily risk of pregnancy for that day, which they can then use to avoid having unprotected sex. The study is being conducted by the Institute for Reproductive Health (IRH) at Georgetown University.

The study will examine the relationship between women's use of the Dot method (both perfect and typical use) and their pregnancy outcomes at the end of the study. The study will also look at several additional secondary outcomes, such as perceived partner support for the method, coital frequency during the fertile time, and intention to continue using the method after study discontinuation, as well as several other variables around the acceptability of conducting an efficacy study via an app.

The study will recruit women who have already downloaded the DOT app on their Android phones. The study will only recruit women who have previously set their intent in the Dot app as "avoid pregnancy" and entered their second period start date into the app. Eligible women will be: between 18 and 39 years old, have not been pregnant or used hormonal contraception in the last 3 months, are sexually active in a relationship with a male partner, and desire to avoid pregnancy for at least one year.

Women who are consented and entered into the study will activate a "research module" within the Dot app. This module is essentially an "overlay" to the DOT app. It does not change the app itself in any way, but provides a data platform for researchers to obtain self-reported data from study participants about their daily sexual history and to collect periodic surveys from participants on topics pertaining to the study primary and secondary outcomes. Women who report pregnancy, or who fail to enter a new cycle start date within the 40-day window allowed by the Dot method, will be contacted and sent urine pregnancy tests, to confirm their pregnancy status. Participants will complete a maximum of 13 menstrual cycles (approximately 1 year) in the study.

ELIGIBILITY:
Inclusion Criteria:

* Have downloaded the Android app and selected to use it for pregnancy prevention and have indicated that they are interested in participating in the study;
* Have provided contact information to learn more about the study or called the call center;
* Are between 18 and 39 at the time of admission;
* Have menstrual cycles between 20-40 days at the time of enrollment
* Are sexually active with a male partner;
* Have not been pregnant or using any hormonal method of family planning within the past three months
* Are willing to install a password or biometric protection on their phone to ensure the confidentiality of their study data; and
* Live in the U.S.

Exclusion Criteria:

Women who do not meet one or more of the inclusion criteria will be excluded from the study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of eligible participants for this study is women who 1) have begun using Dot for pregnancy prevention; 2) entered their second period start date (i.e., have completed one cycle - in whole or in part - of Dot use), and 3) have indicated that their first cycle was 20-40 days long.
Sampling Method: Non-Probability Sample
Enrollment: 718 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Jennings, PhD, Principal Investigator — Institute for Reproductive Health at Georgetown University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li D, Heyer L, Jennings VH, Smith CA, Dunson DB. Personalised estimation of a woman's most fertile days. Eur J Contracept Reprod Health Care. 2016 Aug;21(4):323-8. doi: 10.1080/13625187.2016.1196485. Epub 2016 Jun 14. PMID 27297611
- [Background] Simmons RG, Shattuck DC, Jennings VH. Assessing the Efficacy of an App-Based Method of Family Planning: The Dot Study Protocol. JMIR Res Protoc. 2017 Jan 18;6(1):e5. doi: 10.2196/resprot.6886. PMID 28100441
- [Result] Jennings VH, Haile LT, Simmons RG, Fultz HM, Shattuck D. Estimating six-cycle efficacy of the Dot app for pregnancy prevention. Contraception. 2019 Jan;99(1):52-55. doi: 10.1016/j.contraception.2018.10.002. Epub 2018 Oct 11. PMID 30316782
- [Result] Jennings V, Haile LT, Simmons RG, Spieler J, Shattuck D. Perfect- and typical-use effectiveness of the Dot fertility app over 13 cycles: results from a prospective contraceptive effectiveness trial. Eur J Contracept Reprod Health Care. 2019 Apr;24(2):148-153. doi: 10.1080/13625187.2019.1581164. Epub 2019 Mar 18. PMID 30880509
- [Derived] Shattuck D, Haile LT, Simmons RG. Lessons From the Dot Contraceptive Efficacy Study: Analysis of the Use of Agile Development to Improve Recruitment and Enrollment for mHealth Research. JMIR Mhealth Uhealth. 2018 Apr 20;6(4):e99. doi: 10.2196/mhealth.9661. PMID 29678802

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women Using Dot to Avoid Pregnancy
Started | 718
Completed | 336
Not Completed | 382

BASELINE CHARACTERISTICS:
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 718
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 718
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 718
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethincity: American Indian or Alaska Native | 6
  Race and Ethincity: Asian | 6
  Race and Ethincity: Native Hawaiian or Other Pacific Islander | 2
  Race and Ethincity: Hispanic or Latino | 118
  Race and Ethincity: Black or African American | 134
  Race and Ethincity: White | 396
  Race and Ethincity: Other | 35
  Race and Ethincity: Unknown or Not Reported | 21
Region of Enrollment [Number; unit: participants]
  United States | 718

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rates
Description: Pregnancy rates during perfect and typical use of the Dynamic Optimal Timing method to avoid pregnancy in a way directly comparable to the approach used in recent family planning effectiveness studies
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 718
Participants | 25

2. Secondary Outcome: Intent to Continue Using the Method at Study Completion
Description: 46.8% of women reported on their 13th cycle that they intend to keep using Dot to prevent pregnancy.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 718
Participants | 336

3. Secondary Outcome: Perceived Partner Support
Description: 687 out of 718 women completed the survey where we asked about perceived partner support. The survey was not mandatory and some women did not complete the study or exited the study prior to its administration.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 687
Participants | 609

4. Secondary Outcome: User Acceptability of App-based, Self-reported Data Collection
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 718
Participants | 682

5. Secondary Outcome: User Perceived Impact of the Dot App
Description: The Dot app has increased my awareness of the importance of knowing my fertile window, in order to prevent pregnancy
Time Frame: 1 year
Population: Users who took the 10-month follow-up survey
Measure: Count of Participants; unit: Participants
Arm/Group | Women Using Dot to Avoid Pregnancy
Number analyzed (Participants) | 371
Participants | 319

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Women Using Dot to Avoid Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/718
Serious Adverse Events (participants affected / at risk) | 0/718
Other Adverse Events (participants affected / at risk) | 0/718

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-01-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT02833922/Prot_000.pdf